CLINICAL TRIAL: NCT07326293
Title: The Effectiveness of Oxygen Reserve Index in Early Detection of Desaturation in Geriatric Patients Scheduled for Oncological Surgery; a Prospective, Observational Study.
Brief Title: The Effectiveness of Oxygen Reserve Index in Early Detection of Desaturation in Geriatric Patients Scheduled for Oncological Surgery
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-24-8204
Record Dates: First submitted 2025-12-18; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Desaturation; Apnea, Hypoxia; Oxygen Reserve Index
Keywords: oxygen reserve indec; geriatric; desaturation
MeSH Terms: conditions — Apnea; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study aims to evaluate the relationship between the Oxygen Reserve Index (ORI) and tolerable apnea time in geriatric patients undergoing elective oncologic surgery under general anesthesia.

Patients aged 65 years and older will be monitored using standard anesthesia monitoring and Masimo Rainbow SET® Pulse CO-Oximetry during anesthesia induction and tracheal intubation.

Tolerable apnea time will be defined as the duration from the end of ventilation after intubation to a decrease in peripheral oxygen saturation (SpO₂) to 94%.

The primary objective is to assess the association between ORI warning time and tolerable apnea time. Secondary objectives include evaluating the association between ORI values, arterial blood gas parameters at predefined time points, and the Clinical Frailty Scale.

DETAILED DESCRIPTION:
This study is a prospective, observational study. Patients aged 65 years and older who are scheduled for elective oncologic surgery at Ankara Bilkent City Hospital will be included. In all patients, the Clinical Frailty Scale will be routinely assessed during the preoperative period.

In this study, tolerable apnea time will be defined as the time until peripheral oxygen saturation (SpO₂), measured by pulse oximetry, decreases to 94%. Although SpO₂ values of 90% and above have been accepted in the literature, the World Health Organization defines normal SpO₂ as 95% and above and considers values of 94% and below as an indication for treatment.

The Oxygen Reserve Index (ORI) ranges from 0 to 1, and the ORI alarm value triggered by the device due to a downward trend will be recorded. ORI is a dimensionless index ranging from 1 (high oxygen reserve) to 0 (no oxygen reserve), which is measured by optically detecting changes in venous oxygen saturation (SvO₂) after arterial oxygen saturation (SpO₂) reaches 100%. ORI is measured using a multi-wavelength pulse co-oximeter placed on a fingertip.

In addition to routine anesthesia monitoring, including electrocardiography, pulse oximetry, and hemodynamic monitoring, patients will also be monitored using Masimo Rainbow SET® Pulse CO-Oximetry. Due to the oncologic nature of the surgeries and the associated risk of bleeding, close hemodynamic monitoring is required; therefore, invasive arterial blood pressure monitoring will be established in all patients before anesthesia induction.

All patients will be preoxygenated with 100% oxygen for 3 minutes. After establishing intravenous access, anesthesia induction will be performed using intravenous propofol at a dose of 2 mg/kg and fentanyl at a dose of 1 µg/kg. Neuromuscular blockade will be achieved with rocuronium at a dose of 0.6 mg/kg.

All patients will be intubated by an experienced anesthesiologist using a videolaryngoscope. Oxygen Reserve Index (ORI) and peripheral oxygen saturation (SpO₂) values will be recorded, and arterial blood gas analyses will be performed at five predefined time points: baseline (initial values), after 3 minutes of preoxygenation, after 2 minutes of bag-mask ventilation following intubation, during apnea when SpO₂ decreases to 94% without ventilation, and after 2 minutes of ventilation with 100% oxygen.

ORI warning time will be defined as the interval from the onset of the ORI alarm to the decrease of SpO₂ to 94%. SpO₂ warning time will be defined as the duration of the decrease in SpO₂ from 97% to 94%.

ELIGIBILITY:
Inclusion criteria for the files/records/materials to be included in the study:

Records of patients aged 65 years and older, classified as ASA physical status I-III, who are scheduled for elective oncologic surgery.

Exclusion criteria for the files/records/materials to be included in the study:

Records of patients with advanced coronary artery disease; advanced heart failure and/or valvular heart disease; carotid artery stenosis; left ventricular ejection fraction below 30%; rapid atrial fibrillation; body mass index (BMI) greater than 35 kg/m²; anticipated difficult airway; advanced-stage malignancy; or dementia.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Study Population: It will be studied in patients over the age of 65.
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-02-16 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the association between Oxygen Reserve Index (ORI) warning time and tolerable apnea time. ORI warning time is defined as the time interval from the onset of the ORI alarm triggered by a downward trend to the decrease of per | Peri-induction period at predefined time points baseline; after 3 minutes of preoxygenation; after 2 minutes of bag-mask ventilation following intubation; during apnea at SpO₂ 94%; and after 2 minutes of ventilation with 100% oxygen
  The primary outcome measure is the association between Oxygen Reserve Index (ORI) warning time and tolerable apnea time.
  ORI warning time is defined as the time interval from the onset of the ORI alarm triggered by a downward trend to the decrease of peripheral oxygen saturation (SpO₂) to 94%.
  Tolerable apnea time is defined as the duration from the end of ventilation after tracheal intubation to the decrease of SpO₂ to 94%.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)